CLINICAL TRIAL: NCT02343965
Title: The Impact of the Practice of Touch-massage on the Anxiety of Patients With Hematological Disorders Hospitalized in a Protective Environment, a Randomized, Controlled Study
Acronym: TANDHEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC14_0202
Record Dates: First submitted 2015-01-12; First posted 2015-01-22 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Hematologic Diseases
Keywords: Touch-massage; anxiety; leukemia; haematology; cancerology; supportive care; complementary therapy
MeSH Terms: conditions — Hematologic Diseases; Anxiety Disorders; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Touch-massage group (Experimental): Patient receive 3 sessions of touch-massage (the duration of a session of touch massage is 15 minutes) ,once a week, for 3 weeks
  Interventions: Other: Touch-massage
- without touch-massage group (No Intervention)

INTERVENTIONS:
Other: Touch-massage
  Arms: Touch-massage group

SUMMARY:
Each year, 17000 cases of severe hematological diseases are diagnosed in France, with more than 6,000 of these requiring hospitalization in a protective, sterile environment. New methods, such as touch massage, have emerged in response to anxiety symptoms observed in patients in such sterile and isolated surroundings. We hypothesize that during the period of isolation, touch massage becomes a nursing care which can help the patient.

DETAILED DESCRIPTION:
Patients with hematologic diseases (leukaemia, myeloma, lymphoma) hospitalized in a sterile area of a hematology unit for at least 3 weeks 18 to 65 years female or male Not having met the nurse, who is providing the touch-massage

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic diseases (leukaemia, Myeloma, lymphoma) hospitalized in a sterile area of a hematology unit for at least 3 weeks
* 18 to 65 years
* Female or male
* Not having met the nurse, who is providing the touch-massage

Exclusion Criteria:

* Allergy to sweet almond oil
* Injury to the skin, at the back and / or arms and / or hands
* Cognitive impairment and / or preventing psychiatric responses to interviews and / or questionnaires
* Physical inability to take sitting in an ergonomic chair for the conduct of touch massage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Impact of touch-massage practice on patients' anxiety state, as measured by the anxiety-state questionnaire (Spielberger, CD et al, 1983) to assess the predisposition to anxiety. | 3 weeks
  Each patient will complete the anxiety-state questionnaire (Spielberger, CD et al, 1983) to assess the predisposition to anxiety.
  The evolution of patient anxiety is calculated from the six scores of the anxiety-state scale administered before and after each of the 3 sessions of touch-massageusing the trait anxiety scale score.

SECONDARY OUTCOMES:
Evolution of Self Esteem, as measured by the self-esteem questionnaire | 3 weeks
  Each patient will complete the self-esteem questionnaire before the first and after the final session of touch-massage .
Evolution of anxiety, measured by the the anxiety-state questionnaire (Spielberger, CD et al, 1983) | 3 weeks
  Each patient will complete the anxiety-state questionnaire (Spielberger, CD et al, 1983) to assess the predisposition to anxiety.
  The evolution of patient anxiety is calculated from the six scores of the anxiety-state scale administered before and after each of the 3 sessions of touch-massageusing the trait anxiety scale score.
Evolution of anxiety | 3 weeks
  Quantitative Analysis about 2 interviews recorded.In order to complement and enrich the quantitative data, two interviews will be conducted with patients receiving send the touch-massage. The data collected will be subjected to a thematic content analysis.

REFERENCES:
- [Derived] Simon A, Nizard JJ, Chevalier P, Le Gouill S, Rulleau T, Planche L, Evin A. Impact of the practice of touch-massage(R) by a nurse on the anxiety of patients with hematological disorders hospitalized in a sterile environment, a randomized, controlled study. BMC Complement Med Ther. 2024 Jan 2;24(1):1. doi: 10.1186/s12906-023-04302-3. PMID 38167315